CLINICAL TRIAL: NCT03399994
Title: A Randomized Clinical Trial of Abluminus DES+ Sirolimus Eluting Stent Versus Everolimus-eluting DES for Percutaneous Coronary Intervention in Patients With Diabetes Mellitus: an Investigator-initiated Pilot Study
Brief Title: Clinical Trial of Abluminus DES+ Sirolimus Eluting Stent Versus Everolimus-eluting DES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Evidence per Attività e Ricerche Cardiovascolari ONLUS (Other)
Collaborators: Mediolanum Cardio Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABILITY
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease; Diabetes
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized multi-centre controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: The members of the Event Adjudication Committee will be blinded to the patient assignment. All medical records, source documentation and event information collected for the adjudication process will be blinded to treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABLUMINUS DES+ (Experimental): device implantation during coronary angioplasty
  Interventions: Device: device implantation during coronary angioplasty
- Everolimus-eluting DES (Active Comparator): device implantation during coronary angioplasty
  Interventions: Device: device implantation during coronary angioplasty

INTERVENTIONS:
Device: device implantation during coronary angioplasty — device implantation during coronary angioplasty

SUMMARY:
The objective of the study is to compare angiographic and clinical performance of Abluminus DES+ versus Everolimus-eluting DES in patients with diabetes mellitus.

DETAILED DESCRIPTION:
The present clinical investigation is designed as a prospective, multicentre, national, randomized, open label, 2-arm parallel group, pilot trial comparing Abluminus DES+ versus Everolimus-eluting DES on Late Lumen Loss and clinical outcomes in diabetic patients undergoing Percutaneous Coronary Intervention.

A total of 165 patients will be recruited and randomized in the two groups in a 2:1 ratio at up to 6-8 Italian sites.

After index procedure, patients will be followed up by angiographic follow-up at 9 months and clinical follow-up at 12 months.

The study design is open label, since it is not possible to blind the investigators as to the stent type. However the members of the Event Adjudication Committee will be blinded to the patient. assignment. All medical records, source documentation and event information collected for the adjudication process will be blinded to treatment assignment.

In addition the primary endpoint will be independently evaluated by the Core-Lab which will be blinded as to group assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18
2. Diabetes mellitus
3. Documented CAD: stable or unstable angina, Non-ST segment MI, silent ischemia or positive functional study
4. PCI considered appropriate and feasible
5. Culprit de novo lesion in a native coronary artery with significant stenosis (>50% by visual estimate) eligible for stent implantation (no limitation on the number of treated lesions, vessel and lesion length);
6. Patient provides written informed consent
7. Patient agrees to all required follow-up procedures and visits.
8. Target lesion suitable for PCI with DES diameter between 2.5 and 4.0 mm.

Exclusion Criteria:

1. The patient has a known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, ticlopidine, sirolimus, everolimus, and/or contrast media (patients with documented sensitivity to contrast which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Patients with true anaphylaxis to prior contrast media, however, should not be enrolled);
2. Any contraindication to the implant of the Abluminus DES+
3. Subject is pregnant, nursing, or is a woman of child-bearing potential who is not surgically sterile, 2 years postmenopausal, or does not consistently use effective methods of contraception;;
4. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions;
5. Previous coronary intervention on target vessel in the 3-months prior to enrollment;
6. Non-cardiac co-morbid conditions with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment);
7. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period;
8. Previously documented left ventricular ejection fraction (LVEF) <30%;
9. Evident cardiogenic shock before randomization;
10. Patients with left main stem stenosis (>50% by visual estimate);
11. In-stent restenosis;
12. ST-segment elevation MI;
13. Chronic total occlusion.
14. Culprit lesion to a Saphenous Vein graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
In-stent neointimal volume | 9-month follow-up
  In-stent neointimal volume, measured with OCT, following PCI with Abluminus DES+ compared with in-stent neointimal volume following PCI with Everolimus-eluting DES.

SECONDARY OUTCOMES:
Neointimal area | 9-month follow-up
  Neointimal area, calculated at the site of minimal lumen area measured with OCT.
Target Lesion Failure | 12 months
  This will be a composite of cardiac death, target-vessel MI, and clinically indicated TLR
Stent thrombosis | 12 months
  This is defined according to classification proposed by the Academic Research Consortium
Cardiac death | 12 months
  Any death due to proximate cardiac cause (eg, MI, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure-related deaths, including those related to concomitant treatment, will be classified as cardiac death.
Target vessel myocardial infarction | 12 months
  Any MI that, irrespective of the time after the index procedure, is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause33 Type of acute MI is classified according to the Joint ESC/ACCF/AHA/ WHF Joint Task Force for the Universal Definition of Myocardial Infarction
Target lesion revascularization | 12 months
  repeat revascularization will be defined as any repeat PCI or new coronary artery bypass graft (CABG) surgery within the first year post-PCI.
Device success at 24 hours | 24 hours
  deployment of the assigned stents without system failure or device-related complication
Lesion success | 24 hours
  Attainment of <50% residual stenosis of the target lesion using post-PCI
Procedural success | 24 hours
  Lesion success without the occurrence of Major Adverse Cardiac Events during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, MD, Study Director — Ospedale San Raffaele; Azeem Latib, MD, Principal Investigator — Ospedale San Raffaele
Locations (6):
- Italy (6):
  - Ospedale San Raffaele, Miano, Milano
  - Ospedale Humanitas, Rozzano, Milano
  - Policlinico San Donato, San Donato Milanese, Milano
  - Azienda Ospedaliero Universitaria Policlinico Federico II, Napoli
  - Policlinico S. Matteo, Pavia
  - Ospedale San Pietro, Fatebenefratelli, Roma

IPD SHARING:
Plan to Share IPD: No